CLINICAL TRIAL: NCT03080038
Title: SQUEEZE Trial: A Trial to Determine Whether Septic Shock Reversal is Quicker in Pediatric Patients Randomized to an Early Goal Directed Fluid Sparing Strategy vs. Usual Care
Acronym: SQUEEZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Critical Care Trials Group (Other); Pediatric Emergency Research Canada (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Blood Services (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Melissa Parker, Associate Professor of Pediatrics, McMaster University; Staff Physician, McMaster Children's Hospital, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0833
Record Dates: First submitted 2017-02-28; First posted 2017-03-15 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Septic Shock
Keywords: Sepsis; Shock; Septic Shock; Fluid Therapy; Resuscitation; Pediatrics; Emergency Medicine; Critical Care
MeSH Terms: conditions — Shock, Septic; Sepsis; Shock

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Resuscitation Strategy (No Intervention): Decisions regarding the IV/IO administration of isotonic fluid boluses and/or the initiation and escalation of vasoactive medication infusions are left to the discretion of the treating physician and medical team. We ask that vasoactive medications not be initiated until at least 60 mL/kg (3 litres for children ≥ 50 kg) of isotonic fluid bolus therapy has been administered. The treating physician and medical team are advised to follow ACCM guidelines for the resuscitation of neonatal and pediatric septic shock and to target ACCM recommended therapeutic endpoints.
- Fluid Sparing Resuscitation Strategy (Experimental): The treating physician and medical team are advised to follow the assigned Fluid Sparing Resuscitation Strategy to guide decisions regarding the IV/IO administration of further isotonic fluid boluses, and the timing of initiation and escalation of vasoactive medication infusions to target the therapeutic endpoints recommended in the ACCM guidelines for the resuscitation of neonatal and pediatric septic shock.
  Interventions: Other: Fluid Sparing Resuscitation Strategy

INTERVENTIONS:
Other: Fluid Sparing Resuscitation Strategy — Tier 1: Initiate IV/IO vasoactive medication infusion support immediately. Further IV/IO isotonic fluid bolus therapy [crystalloid (0.9% Normal Saline or Ringers Lactate) or colloid (5% Albumin)] should be avoided; small volume isotonic fluid boluses [5-10 mL/kg (250-500 mL for participants ≥ 50 kg)] may be provided if required due to A. Clinically unacceptable delay in ability to initiate vasoactive medication infusion(s) and/or 2. Documented intravascular hypovolemia.
  Tier 2: Vasoactive medication(s) should be preferentially titrated/escalated to achieve recommended ACCM hemodynamic goals. Further IV/IO isotonic fluid bolus therapy [crystalloid (0.9% Normal Saline or Ringers Lactate) or colloid (5% Albumin)] should be avoided; small volume isotonic fluid boluses [5-10 mL/kg (250-500 mL for participants ≥ 50 kg)] may be provided if required due to A. Documented intravascular hypovolemia.
  Intervention end: Patient is free from vasoactive medication support and shock is reversed.
  Arms: Fluid Sparing Resuscitation Strategy

SUMMARY:
The purpose of the SQUEEZE Trial is to determine which fluid resuscitation strategy results in the best outcomes for children treated for suspected or confirmed septic shock. In this study, eligible children will be randomized to either the 'Usual Care Arm' or the 'Fluid Sparing Arm'. Children will receive treatment according to current ACCM Septic Shock Resuscitation Guidelines, with the assigned resuscitation strategy used to guide administration of further fluid boluses as well as the timing of initiation and escalation of vasoactive medications to achieve ACCM recommended hemodynamic targets.

DETAILED DESCRIPTION:
Please see published pilot trial protocol for more information about the SQUEEZE Trial and rationale for this study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for 1 and 3 must be answered YES to be eligible for study.

* Age 29 days to less than 18 years of age
* Patient has Persistent Signs of Shock including one or more of the following:

  * Vasoactive Medication Dependence
  * Hypotension (Systolic Blood Pressure and/or Mean Blood Pressure less than the 5th percentile for age)
  * Abnormal Perfusion (2 or more of: abnormal capillary refill, tachycardia, decreased level of consciousness, decreased urine output)
* Suspected or Confirmed Septic Shock (Shock due to Suspected or Confirmed Infectious Cause)
* Patient has received initial fluid resuscitation of: Minimum of 40 mL/kg of isotonic crystalloid (0.9% Normal Saline and/or Ringer's Lactate) and/or colloid (5% albumin) as fluid boluses within the previous 6 hours for patients weighing less than 50 kg, OR Minimum of 2 litres (2000 mL) of isotonic crystalloid (0.9% Normal Saline and/or Ringer's Lactate) and/or colloid (5% albumin) as fluid boluses within the previous 6 hours for patients weighing 50 kg or more.
* Patient has Fluid Refractory Septic Shock as defined by the Presence of all of 2a, 2b, and 2c.

Exclusion Criteria:

* Patient admitted to the Neonatal Intensive Care Unit (NICU)
* Patient requiring resuscitation in the Operating Room (OR) or Post-Anesthetic Care Unit (PACU)
* Full active resuscitative treatment not within the goals of care
* Shock Secondary to Cause other than Sepsis (i.e. obvious signs of cardiogenic shock, anaphylactic shock, hemorrhagic shock, spinal shock)
* Previous enrolment in this trial, where known by the research team

Ages: 29 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 406 (Actual)
Dates: Start 2017-03-06 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Difference in time to shock reversal | This outcome can be ascertained typically within 14 days of randomization
  Difference (in hours) in time to shock reversal between the two study groups. Not available where death occurs while still in shock, or if the patient is placed on mechanical circulatory support for refractory shock.

SECONDARY OUTCOMES:
Measures of Organ Dysfunction - Pediatric logistic organ dysfunction score | 28 days
  Pediatric logistic organ dysfunction score
Measures of Organ Dysfunction - Acute Kidney Injury | 28 days
  Acute Kidney Injury
Measures of Organ Dysfunction - Ventilator Free Days | 28 days
  Ventilator Free Days
Complications possibly attributable to fluid overload or third spacing of fluids - Soft tissue edema | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Soft tissue edema
Complications possibly attributable to fluid overload or third spacing of fluids - Pulmonary edema | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Pulmonary edema
Complications possibly attributable to fluid overload or third spacing of fluids - Pleural effusion requiring drainage | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Pleural effusion requiring drainage
Complications possibly attributable to fluid overload or third spacing of fluids - Abdominal Compartment Syndrome | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Abdominal Compartment Syndrome
Complications possibly attributable to fluid overload or third spacing of fluids - Diuretic Exposure | From randomization until 7 days after shock is reversed
  Diuretic Exposure
Complications possibly attributable to inotrope/vasopressor use - Clinical signs of digital tissue schema | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Clinical signs of digital tissue schema
Complications possibly attributable to inotrope/vasopressor use - Digital ischemia requiring revision amputation | 90 days
  Digital ischemia requiring revision amputation
Complications possibly attributable to inotrope/vasopressor use - Clinical signs of compromised bowel perfusion | From randomization until 7 days after shock is reversed
  Clinical signs of compromised bowel perfusion
Critical Care Treatments as binary measurement yes/no | Intervention Period (from randomization until shock is reversed; typically within 14 days)
  Critical care treatments performed during intervention period.
Paediatric Intensive Care Unit Length of Stay | Up to 90 days
  Paediatric Intensive Care Unit Length of Stay
Hospital Length of Stay | Up to 90 days
  Hospital Length of Stay
Mortality Measures | 28-, 90- day, hospital mortality
  Death
Health Service Outcomes - Paediatric Intensive Care Unit Admission Rate | 28 days
  Paediatric Intensive Care Unit Admission Rate

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Parker, MD, MSc, Principal Investigator — McMaster Children's Hospital and McMaster University
Locations (8):
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Sickkids, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The final trial data set will be made public.

REFERENCES:
- [Background] Parker MJ, Thabane L, Fox-Robichaud A, Liaw P, Choong K; Canadian Critical Care Trials Group and the Canadian Critical Care Translational Biology Group. A trial to determine whether septic shock-reversal is quicker in pediatric patients randomized to an early goal-directed fluid-sparing strategy versus usual care (SQUEEZE): study protocol for a pilot randomized controlled trial. Trials. 2016 Nov 22;17(1):556. doi: 10.1186/s13063-016-1689-2. PMID 27876084
- [Derived] Parker MJ, Foster G, Fox-Robichaud A, Choong K, Mbuagbaw L, Thabane L; With the SQUEEZE Trial Steering Committee and on behalf of the SQUEEZE Trial Investigators, the Canadian Critical Care Trials Group, Pediatric Emergency Research Canada, and the Canadian Critical Care Translational Biology Group. Statistical analysis plan for the SQUEEZE trial: A trial to determine whether septic shock reversal is quicker in pediatric patients randomized to an early goal-directed fluid-sparing strategy vs. usual care (SQUEEZE). Crit Care Resusc. 2024 Jun 22;26(2):123-134. doi: 10.1016/j.ccrj.2024.02.002. eCollection 2024 Jun. PMID 39072232
- [Derived] Parker MJ. What Goes Up, Must Go Down? Pediatr Crit Care Med. 2018 Jun;19(6):579-581. doi: 10.1097/PCC.0000000000001543. No abstract available. PMID 29863640
- See also: A trial to determine whether septic shock-reversal is quicker in pediatric patients randomized to an early goal-directed fluid-sparing strategy versus usual care (SQUEEZE): study protocol for a pilot randomized controlled trial — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-016-1689-2